CLINICAL TRIAL: NCT05092516
Title: Home-based Transcranial Direct Current Stimulation (tDCS) for Treatment of Cognitive Post-acute Sequelae of COVID-19 (PASC)
Brief Title: Home-based Brain Stimulation Treatment for Post-acute Sequelae of COVID-19 (PASC)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Hamdi Eryilmaz, PhD, Assistant Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021P002953
Record Dates: First submitted 2021-10-21; First posted 2021-10-25 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Dysexecutive Syndrome; Post-Acute Sequelae of COVID-19
Keywords: Transcranial Direct Current Stimulation; EEG; Sustained attention
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Active tDCS (Experimental): This group will receive daily active stimulation (2 mA) to the left dorsolateral prefrontal cortex for 4 weeks through a home-based tDCS device in remotely-supervised 30-min sessions.
  Interventions: Device: Active tDCS
- Sham tDCS (Sham Comparator): This group will receive daily sham stimulation to the left dorsolateral prefrontal cortex for 4 weeks through a home-based tDCS device in remotely-supervised 30-min sessions.
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Active tDCS — 2 mA of anodal stimulation will be applied to the left prefrontal cortex over the F3 electrode based on the International 10-10 EEG system.
  Arms: Active tDCS
Device: Sham tDCS — Sham stimulation will be applied to the left prefrontal cortex over the F3 electrode.
  Arms: Sham tDCS

SUMMARY:
The main goal of this study is to improve dysexecutive symptoms (e.g., sustained attention, processing speed) in patients exhibiting post-acute sequelae of COVID-19 (PASC) through home-based transcranial direct current stimulation (tDCS), a noninvasive method that uses low intensity electric currents delivered to the brain through stimulation electrodes on the scalp.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* A diagnosis of PASC as indicated by past COVID-19 infection, and persistent symptoms, including 'brain fog', confusion, short-term memory deficits, trouble concentrating, delirium, difficulties in multitasking.

Exclusion Criteria:

* History of epilepsy
* Metallic implants in the head and neck,
* Brain stimulators
* Pacemakers
* Pregnancy
* Active substance dependence (except for tobacco)
* Premorbid major neurological illness
* Severe mental illness (e.g., bipolar disorder, schizophrenia)
* Attention Deficit Hyperactivity Disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-06-07 (Actual); Primary Completion 2025-03-13 (Actual); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Change in inhibitory control | 8 weeks
  Performance during the incongruent trials of the Eriksen Flanker Task will be assessed at four time points before, during, and after the 4-week intervention.
Change in processing speed | 8 weeks
  Reaction time during the incongruent trials of the Eriksen Flanker Task will be assessed at four time points before, during, and after the 4-week intervention.
Change in EEG P300 event-related potential | 8 weeks
  EEG P300 amplitudes time-locked to the incongruent trials of the Eriksen Flanker Task will be assessed at four time points before, during, and after the 4-week intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No